CLINICAL TRIAL: NCT00148057
Title: An Explanatory Clinical Trial of Breast Cancer Prevention
Brief Title: Diet and Breast Cancer Prevention Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Breast Cancer Research Alliance (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01-0428-C; 14177
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2005-09-07 (Estimated); Status verified 2005-08

CONDITIONS: Breast Cancer
Keywords: Diet; Dietary fat; Breast cancer; Prevention
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet, Fat-Restricted

INTERVENTIONS:
Behavioral: Low-fat diet

SUMMARY:
This randomized controlled trial tests the hypothesis that a reduction in intake of dietary fat will reduce the incidence of breast cancer. Women with more than 50% of the breast occupied by dense tissue on a mammogram have been recruited and allocated by a random (ie chance) process, to an intervention or control group. The intervention group has been taught how to reduce their fat intake to a target of 15% of total calories, while the control group continued their usual consumption of fat. Both groups have then been followed for at least 7 years and the number who develop breast cancer in each group will be compared

DETAILED DESCRIPTION:
The long term goal of this trial is to determine if intervention in subjects with extensive mammographic densities (a risk factor for breast cancer) with a low fat-high carbohydrate diet will reduce the incidence of breast cancer by 37%. We propose to meet this goal by carrying out a randomized multi-centre trial of dietary intervention in subjects at increased risk of breast cancer that is now in progress.

The method used is to recruit subjects with extensive mammographic densities and enrol them in a randomized trial in which they receive one of two kinds of dietary counselling. A control group receives general advice about nutrition but is not counselled to change their intake of dietary fat or carbohydrate, and an intervention group is given intensive counselling to reduce their intake of total fat to a target of 15% of calories and increase intake of carbohydrate to maintain intake of total calories.

Recruitment to this trial has been in progress in Toronto, Hamilton, London and Windsor since 1991, and in Vancouver since 1994, and all of the 4,615 subjects required for the trial were recruited by November 1998.

The trial is explanatory in that it seeks to determine if there is a biological effect of dietary fat reduction in terms of a reduction in breast cancer incidence. To meet this goal we will select as participants highly motivated subjects who are at increased risk of breast cancer, provide them with a high level of assistance in making a dietary alteration, follow them carefully to ensure the correct identification of subjects who develop breast cancer, and analyse the results both according to intention to treat and dietary compliance. This trial does not attempt to assess directly the possible effects of dietary counselling on the health of the general public.

II Specific Aims

1. To recruit 4,615 Canadian women with extensive mammographic density and to enrol them in a randomized trial of dietary fat reduction and follow up until 2006.
2. To compare in the control and intervention groups of this trial the incidence of breast cancers, as well as other histological changes in the breast tissue of patients undergoing surgical biopsy of the breast.
3. To determine if a reduction in dietary fat intake will reduce either the proportion of the breast area occupied by radiological signs of density or the total quantity of density.

ELIGIBILITY:
Inclusion Criteria:

1. A mammogram with at least 50% of the breast area occupied by radiological signs of density.
2. Aged more than 30 years and less than 65 years.
3. Body Mass Index >19 and <27.
4. Resident within easy commuting distance of a participating centre. -

Exclusion Criteria:

1. A previous history of cancer (excluding non-melanomatous skin cancer).
2. Pregnant (or planning to be) or breast feeding.
3. On a medically prescribed diet for any reason.
4. Habitually (ie. 4 or more times per week) eats more than one meal a day in a restaurant.
5. Previous mammoplasty, either reduction or augmentation.
6. Previous or present treatment for the reduction of blood lipids.
7. Proposed breast biopsy as a result of the initial clinical and/or mammographic examination, until such time as the biopsy has been carried out and is known to be benign

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4695
Dates: Start 1988-01; Study Completion 2005-12

PRIMARY OUTCOMES:
Breast cancer

SECONDARY OUTCOMES:
Other cancers
Benign breast disease

CONTACTS AND LOCATIONS:
Overall Officials: Norman F Boyd, MD, DSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hidaka BH, Kimler BF, Fabian CJ, Carlson SE. An empirically derived dietary pattern associated with breast cancer risk is validated in a nested case-control cohort from a randomized primary prevention trial. Clin Nutr ESPEN. 2017 Feb;17:8-17. doi: 10.1016/j.clnesp.2016.10.008. Epub 2016 Nov 23. PMID 28361752
- [Derived] Martin LJ, Huszti E, Connelly PW, Greenberg CV, Minkin S, Boyd NF. RE: Serum Lipids, Lipoproteins, and Risk of Breast Cancer: A Nested Case-Control Study Using Multiple Time Points. J Natl Cancer Inst. 2016 May 18;108(8):djw126. doi: 10.1093/jnci/djw126. Print 2016 Aug. No abstract available. PMID 27193584
- [Derived] Martin LJ, Li Q, Melnichouk O, Greenberg C, Minkin S, Hislop G, Boyd NF. A randomized trial of dietary intervention for breast cancer prevention. Cancer Res. 2011 Jan 1;71(1):123-33. doi: 10.1158/0008-5472.CAN-10-1436. PMID 21199800